CLINICAL TRIAL: NCT03357757
Title: The LATENT Trial: Lytic Activation To Enhance Neoantigen-directed Therapy A Study to Evaluate the Feasibility and Efficacy of the Combined Use of Avelumab With Valproic Acid for the Treatment of Virus-associated Cancer
Brief Title: Avelumab With Valproic Acid in Virus-associated Cancer
Acronym: LATENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LATENT
Record Dates: First submitted 2017-11-16; First posted 2017-11-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cancer That is Associated With a Chronic Viral Infection; p16 Positive SCCHN; Squamous Cell Carcinoma of the Cervix; p16 Positive Squamous Cell Carcinoma of the Vagina or Vulva; p16 Positive Squamous Cell Carcinoma of the Penis; p16 Positive Squamous Cell Carcinoma of the Anus or Anal Canal; EBER Positive NPC; EBER Positive Hodgkins and Non-hodgkins Lymphona
MeSH Terms: interventions — Valproic Acid; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Avelumab with VPA (Experimental): Valproic Acid (VPA, 12.5 mg/kg) once per day and Avelumab (10 mg/kg IV) every 2 weeks for up to 2 years.
  Interventions: Drug: Valproic Acid; Biological: Avelumab

INTERVENTIONS:
Drug: Valproic Acid — The target serum level for VPA will be between 75 and 100 mcg/mL checked every 2 weeks for the first 6 cycles.
Biological: Avelumab — 10 mg/kg IV

SUMMARY:
Up to 20% of all cancers may be associated with a bacterial or viral infection. In some instances, the infection may be one of the reasons why the cancer developed in the first place. One such example is infection with the human papilloma virus (HPV) and the development of cervical or oral cavity cancer.

A viral infection that is chronic may not cause a person symptoms, and may be able to escape detection by a person's own immune system. One of the medications being studied in this clinical trial (Valproic acid) may be able to unmask a chronic viral infection from a person's own immune system, therefore making the virus susceptible to attack by the immune system. In this study Valproic acid is being combined with an immune therapy, Avelumab. Avelumab is an antibody that targets a person's own immune cells, or lymphocytes. Lymphocytes must be activated to fight infections or cancer, but after activation they are deactivated. Avelumab prevents the deactivation of a lymphocyte, in effect "turning off the off-switch." This leads to a re-energizing of a person's immune system, hopefully leading to an attack by the immune system on a person's cancer.

Avelumab is known to be an effective treatment for a variety of cancers, although it has not yet been tested in all cancers. By combining Valproic acid, a treatment which targets the virus that contributed to the development of this type of cancer with Avelumab the investigators hope to enhance the ability of Avelumab to restore the body's own immune defense against the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Patients with the following histologically confirmed diagnoses will be eligible for enrolment: p16 positive SCCHN; squamous cell carcinoma of the cervix; p16 positive squamous cell carcinoma of the vagina or vulva; p16 positive squamous cell carcinoma of the penis; p16 positive squamous cell carcinoma of the anus or anal canal; EBER positive NPC; EBER positive Hodgkins and non-hodgkins lymphoma.
* Note: patients with p16 positive SCC of unknown primary origin meeting the minimum life expectancy and performance status requirements will also be eligible for enrollment, as the majority of these patients may be assumed to represent HPV-associated disease.
* Patients must be capable of providing consent to enrolment and treatment.
* Patients with a performance status of ECOG 0-1(51) will be eligible for enrolment (see appendix 1).
* Measurable disease must be present according to irRECIST criteria(50).
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening.
* Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 60 days after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
* Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 120 days after the last dose of study drug.
* Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
* The following adequate organ function laboratory values must be met:
* Hematological:

  * Absolute neutrophil count (ANC) >1.5 x109/L
  * Platelet count >100 x109/L
  * Hemoglobin >9 g/dL (may have been transfused)
* Renal:

  o Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
* Hepatic:

  * Total serum bilirubin <1.5x ULN
  * AST and ALT <2.5x ULN (or ≤ 5 x ULN for subjects with documented metastatic disease to the liver)
  * Serum albumin > 25 g/L
* Coagulation:

  * International Normalized Ratio (INR) <1.5x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
  * Activated Partial Thromboplastin Time (aPTT) <1.5x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)

Exclusion Criteria:

* History of pneumonitis requiring treatment with steroids.
* History of interstitial lung disease.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* History of another malignancy or a concurrent malignancy;
* Exceptions include patients who have been disease-free for 5 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
* Active brain metastases or leptomeningeal disease.
* Patients with treated brain metastases that are stable for 6 weeks will be eligible for enrolment.
* Diagnosis of immunodeficiency.
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Prior organ transplantation including allogenic stem-cell transplantation.
* Known history of human immunodeficiency virus (HIV).
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Patients with hyperthyroidism or hypothyroidism but that are stable on hormone replacement will not be excluded.
* Active infection requiring systemic therapy.
* Vaccination within 4 weeks of the first dose of Avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* Patient will not be eligible if the patient is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of Avelumab and VPA | 1 year after enrolment of last patient
  • Assessment of the clinical response rate according to the immune-related RECIST criteria (iRECIST)
Proportion of subjects who complete 4 doses of Avelumab in combination with VPA | 1 year after enrolment of last patient
  • Feasibility analysis, defined as the proportion of subjects who complete 4 doses of Avelumab in combination with VPA over the total duration of the study.

SECONDARY OUTCOMES:
Overall survival | 5 years from final study drug dose
  defined as the time from the date of enrollment to the date of death, whatever the cause.
Progression free survival | 5 years from final study drug dose
  Progression free survival is defined as the time between the date of treatment initiation and the date of disease progression or death (whatever the cause), whichever occurs first.
Number of participants with adverse events | Through study completion, up to 2 years
  • Incidence of adverse events (assessed as the incidence and severity of adverse events, including immune-related adverse events, and the number of discontinuations due to adverse events).
Identify specific virus-associated cancers as candidates for subsequent study | Through study completion, up to 2 years
Measurement of Immuno-score | Through study completion, up to 2 years
  AffymetriX Micro-array (Immuno-score)
Measurement of MHC expression | Through study completion, up to 2 years
Measurement of cell-free tumoral DNA in blood | Through study completion, up to 2 years
Phenotyping of Tumour Infiltrating Lymphocytes | Through study completion, up to 2 years
DNA viral load | Through study completion, up to 2 years
  DNA Quantitative PCR (viral load)
Expression of lytic viral genes | Through study completion, up to 2 years
Cytotoxic T-Lymphocyte immunophenotyping | Through study completion, up to 2 years
T-cell receptor sequencing | Through study completion, up to 2 years
Hsp90 concentration in serum | Through study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Walker, MD PhD FRCPC, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No